CLINICAL TRIAL: NCT00867152
Title: A Phase I, Open Label, Randomized, Three Period, One-way, Two Cohort, Adaptive Crossover Study to Evaluate the Effect of Darunavir/Ritonavir Plus Etravirine and Lopinavir/Ritonavir Plus Etravirine on GSK1349572 Pharmacokinetics in Healthy Adult Subjects (ING112934)
Brief Title: GSK1349572 Drug Interaction With Etravirine and Either Darunavir/Ritonavir or Lopinavir/Ritonavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 112934
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Healthy Volunteer
Keywords: ritonavir; GSK1349572; integrase; lopinavir; darunavir; etravirine
MeSH Terms: interventions — Darunavir; etravirine; Ritonavir; Lopinavir; lopinavir-ritonavir drug combination; dolutegravir

ARMS (2):
- Cohort 2 (Experimental): All subjects will receive GSK1349572 50mg q24h (Treatment A) from Day 1 to Day 5 in Period 1. There will be no washout between treatment Periods 1 and 2. Subjects will receive GSK1349572 50mg q24h and ETV/DRV/RTV 200/600/100mg q12h from Day 1 to Day 14 in Period 2. Day 1 of Period 3 will be approximately 3 weeks after the last dose in Period 2. Subjects will receive GSK1349572 50mg q12h and ETV/DRV/RTV 200/600/100mg q12h from Day 1 to Day 14. Period 3 will not be performed if there is no significant interaction in Period 2.
  Interventions: Drug: Darunavir; Drug: Etravirine; Drug: Ritonavir; Drug: GSK1349572
- Cohort 1 (Experimental): All subjects will receive GSK1349572 50mg q24h (Treatment A) from Day 1 to Day 5 in Period 1. There will be no washout between treatment Periods 1 and 2. Subjects will receive GSK1349572 50mg q24h and ETV/LPV/RTV 200/400/100mg q12h from Day 1 to Day 14 in Period 2. Day 1 of Period 3 will be approximately 3 weeks after the last dose in Period 2. Subjects will receive GSK1349572 50mg q12h and ETV/LPV/RTV 200/400/100mg q12h from Day 1 to Day 14. Period 3 will not be performed if there is no significant interaction in Period 2.
  Interventions: Drug: Etravirine; Drug: Lopinavir/ritonavir; Drug: GSK1349572

INTERVENTIONS:
Drug: Darunavir — Darunavir 600 mg every 12 hours for 14 days in Periods 2 and 3. Period 3 may not be done. Darunavir is approved by the FDA as an HIV medication in the protease inhibitor class.
  Other Names: Prezista
  Arms: Cohort 2
Drug: Etravirine — Etravirine 200 mg every 12 hours for 14 days in Periods 2 and 3. Period 3 may not be done. Etravirine is approved by the FDA as an HIV medication in the non-nucleoside reuptake inhibitor class.
  Other Names: Intelence
Drug: Ritonavir — Ritonavir 100 mg every 12 hours for 14 days in Periods 2 and 3. Period 3 may not be done. Ritonavir is approved by the FDA as an HIV medication in the protease inhibitor class.
  Other Names: Norvir
  Arms: Cohort 2
Drug: Lopinavir/ritonavir — Lopinavir 400 mg and ritonavir 100 mg every 12 hours for 14 days in Periods 2 and 3. Period 3 may not be done. Lopinavir/Ritonavir is approved by the FDA as an HIV medication in the protease inhibitor class.
  Other Names: Kaletra
  Arms: Cohort 1
Drug: GSK1349572 — GSK1349572 50 q24h for 5 days in Period 1 and for 14 days in Period 2. GSK1349572 20 mg q12h for 14 days in Period 3 if Period 3 is done. GSK1349572 is an investigational (not approved by the FDA) HIV medication in the integrase inhibitor class.

SUMMARY:
A Phase I, open label, randomized, three period, one-way, two cohort, adaptive crossover study to evaluate the effect of darunavir/ritonavir plus etravirine and lopinavir/ritonavir plus etravirine on GSK1349572 pharmacokinetics in healthy adult subjects

DETAILED DESCRIPTION:
The study is a three period, randomized, open label study. Approximately 18 healthy subjects will receive GSK1349572 50mg q24h for 5 days (Treatment A) in Period 1. Subjects will then be administered GSK1349572 50mg q24h in combination with either LPV/RTV 400/100 mg q12h and etravirine 200mg q12h (Treatment B, n=9) or DRV/RTV 600/100 mg q12h and etravirine 200mg q12h (Treatment C, n=9) for 14 days in Period 2 followed by a washout period. GSK1349572 PK data will be obtained from Periods 1 and 2 and used to inform decision making on Period 3. If GSK1349572 Cτ is reduced by more than 50% in Period 2 compared to Period 1, subjects will return to the clinic and receive GSK1349572 50mg q12h in combination with ETV and either DRV/RTV or LPV/RTV in Period 3. Safety evaluations and serial PK samples will be collected during each treatment period. A follow-up visit will occur 7-14 days after the last dose of study drug. All doses of study drugs will be taken following a moderate fat meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 65 years of age, inclusive.
* A female subject is eligible to participate if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any female who: Is pre-menopausal with a documented bilateral tubal ligation, bilateral oophorectomy (removal of the ovaries) or hysterectomy, or Is postmenopausal defined as 12 months of spontaneous amenorrhea. A follicle stimulating hormone (FSH) level will be performed to confirm a post-menopausal status. For this study, FSH levels of > 40 MlU/ml is confirmatory. For females on hormone replacement therapy (HRT) and whose menopausal status is in doubt, HRT should be discontinued for 2 weeks and then the subject rescreened, as HRT can suppress FSH.
* Male subjects must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until 14 days after the last dose of study medication.
* Body weight ≥ 50 kg for men and ≥ 45 kg for women and BMI within the range 18.5-31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat is allowed for eligibility determination.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive test for HIV antibody.
* A positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids, and benzodiazepines.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* History of regular use of tobacco or nicotine-containing products within 3 months prior to screening.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* History of sensitivity to any of the study medications, or components thereof including sulfa-containing drugs, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* If heparin is used in during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* History of significant renal or hepatic diseases.
* History/evidence of clinically significant pulmonary disease.
* History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA) or any clinically significant cardiac disease.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy, peptic ulceration, inflammatory bowel disease or pancreatitis should be excluded.
* Serum creatinine values greater than the upper limit of normal. A single repeat is allowed for eligibility determination.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100bpm for male subjects.
* Screening ECG outside protocol limits (a single repeat is allowed for eligibility determination)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Plasma GSK1349572 steady-state AUC(0-τ), Cmax, C0, Cτ, and Cmin following administration of GSK1349572 50mg and following co-administration of GSK1349572 50mg with ETV/LPV/RTV 200/400/100mg or ETV/DRV/RTV 200/600/100mg | 14 days

SECONDARY OUTCOMES:
Safety and tolerability parameters, including adverse event, concurrent medication, clinical laboratory, ECG, and vital signs assessments. | 12 weeks
Plasma ETV PK parameters, including AUC(0-τ), Cmax, and Cmin following co-administration of GSK1349572 50mg q24h (and 50mg q12h if appropriate) and ETV/LPV/RTV 200/400/100mg q12h or ETV/DRV/RTV 200/600/100mg q12h | 14 days
GSK1349572 PK parameters, including, tmax, tmin, CL/F and t½ following administration of GSK1349572 50mg q24h for 5 days and following co-administration of GSK1349572 50mg and ETV/LPV/RTV 200/400/100mg q12h or ETV/DRV/RTV 200/600/100mg | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States